CLINICAL TRIAL: NCT00835653
Title: Efficacy of Median Nerve Block Performed Using Echographic Guidance
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/42
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Orthopedic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with a carpal tunnel syndrome
  Interventions: Procedure: median nerve block
- 2: patients without a carpal tunnel syndrome
  Interventions: Procedure: median nerve block

INTERVENTIONS:
Procedure: median nerve block — median nerve block performed under echographic guidance
  Groups: 1
Procedure: median nerve block — median nerve block performed under echographic guidance
  Groups: 2

SUMMARY:
Observational study of the efficacy of median nerve blocks performed using echographic guidance in patients presenting with or without carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* short surgical procedure (less than 30 minutes) on the hand,
* regional anesthesia at the elbow involving the median nerve.

Exclusion Criteria:

* age less than 18 years,
* pregnant woman
* mental incapacity,
* poor understanding of French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for hand surgery
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
light touch sensibility | 30 minutes following block performance

SECONDARY OUTCOMES:
ice touch sensibility | 30 minutes following block performance
motor block | 30 minutes following block performance
paresthesia | during nerve block procedure
vascular puncture | during nerve block procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (2):
- France (2):
  - Hopital Foch, Suresnes
  - Hôpital Privé de l'Ouest Parisien, Trappes